CLINICAL TRIAL: NCT04214210
Title: The DIALOGUE Study: Using Digital Health to Improve Care for Families With Predisposition to Hereditary Cancer
Brief Title: The DIALOGUE Study: Swiss-Korean Billateral Collaboration
Acronym: DIALOGUE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: Yonsei University (Other); University Hospital, Basel, Switzerland (Other); Hopital du Jura, Delemont, Switzerland (Unknown); Department of Computer Science Yonsei University, Seoul, Korea (Unknown); National Cancer Center, Korea (Other Government); Chungnam National University (Other); Ente Ospedaliero Cantonale, Ticino, Switzerland (Other); Swiss National Science Foundation (Other); Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Geneva (Other); Kantonal Hospital Winterthur, Medical Oncology (Unknown); Kantonal Hospital Fribourg, Breast Center (Unknown); Hirslanden, Grangettes, Geneva (Unknown); Kantonal Hospital Solothurn, Olten (Unknown); Kantonal Hospital Graubunden (Unknown); Kantonal Hospital Wallis, Sion (Unknown); Zurich Breast Center (Unknown)
Responsible Party: Principal Investigator, Maria Katapodi, Professor of Nursing, Department of Clinical Research, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: IZKSZ3_188408 / 1
Record Dates: First submitted 2019-11-03; First posted 2020-01-02 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Hereditary Cancer; Breast Cancer; Ovarian Cancer
Keywords: cascade genetic testing; disclosure of genetic test results; family communication; web-based platform; efficacy; implementation outcomes
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tailored Family Gene Toolkit (Experimental): The tailored FGT will include 5 modules designed to increase knowledge of cancer genetics (1); provide decisional support for genetic testing (2); increase active coping to challenges faced by HBOC families (3); provide a 5-steps, skills-building communication training (4); and provide information about management of hereditary cancer risk (5).
  Messages will involve shallow tailoring (e.g. sex of mutation carrier), and deep tailoring with complex elements of relevance (e.g. coping style). Tailoring will be based on personalization, tailored feedback, and content matching, based on Swiss and Korean languages and legislation, health insurance policy, and cultural values.
  Participants will be asked to complete the 5 modules within 4 weeks after they first engage with the intervention. The 4-week interval will enable learning new information while having time to reflect and act. They will receive email alerts to complete the 5 modules with the URL link directing them to the FGT.
  Interventions: Other: Adapted Family Gene Toolkit
- Targeted intervention (Active Comparator): The comparator will provide targeted information about HBOC and enable sharing genetic test results. The Korean team will define the contents of the comparator that will mimic the structure and function of an existing website, already available in the US. The Korean team will create a translation process protocol, and share this guide for further translations from English into Korean and the three Swiss national languages. Both trial arms the tailored and the targeted platform will be technically implemented in the same system, in order to track access and usage of the platform and provide a user-friendly experience to participants. The Swiss team will also provide the implementation of the comparison website.
  Interventions: Other: Targeted intervention

INTERVENTIONS:
Other: Adapted Family Gene Toolkit — Five web-based modules designed to increase knowledge of cancer genetics (Module 1); provide decisional support for genetic testing (Module 2); increase active coping to common challenges faced by HBOC families (Module 3); provide a five-steps, skills-building communication training (Module 4); increase knowledge about management of hereditary cancer risk based on the most updated recommendations from the National Comprehensive Cancer Network (Module 5).
  Arms: Tailored Family Gene Toolkit
Other: Targeted intervention — The comparison website will provide targeted information about HBOC and enable sharing genetic test results.The Korean team will define the contents of the comparison website that will mimic the structure and function of a website already available in the US. The Korean team will create a translation process protocol, and share this guide for further translations from English into Korean and three Swiss national languages. The tailored and the targeted platform will be technically implemented in the same system, to track access and usage of the platform and provide a user-friendly experience.
  Arms: Targeted intervention

SUMMARY:
In Hereditary Breast and Ovarian Cancer (HBOC) communication of genetic test results with relatives is essential to cascade testing. According to privacy laws those identified with the pathogenic variant have the sole responsibility to share information about test results and implications to relatives. Up to 50% of biological relatives are unaware of relevant genetic information, suggesting that benefits of genetic testing are not communicated effectively. Interventions designed to help mutation carriers communicate with relatives are critical for cascade genetic testing. Technology could play a significant role in facilitating communication and genetic education within HBOC families The investigators will develop a digital health platform for Swiss and Korean HBOC families. The digital platform will be based on the Family Gene Toolkit (FGT), a web-based intervention designed to enhance communication of genetic test results within HBOC families that has been tested for acceptability, usability, and participant satisfaction. The investigators will expand a Swiss research infrastructure to enable future collaborative projects between the two countries.

Specific Aims

1. Develop a digital health platform to support the communication of cancer predisposition in HBOC families, based on linguistic and cultural adaptation methods of the FGT for the Swiss and Korean population
2. Develop the K-CASCADE research infrastructure in Korea by expanding the research infrastructure developed by the CASCADE Consortium in Switzerland
3. Evaluate the efficacy of the digital platform on psychological distress and communication of genetic test results, and knowledge of cancer genetics, coping, and decision making
4. Explore the reach, effectiveness, adoption, implementation, and maintenance of the digital platform The digital platform will be based on the FGT with linguistic adaptation for web and mobile access. Aim 1 will be achieved with focus groups with 20-24 HBOC mutation carriers and relatives and 6-10 providers involved in genetic services. For Aim 2, a Korean database of HBOC families (K-CASCADE) will be based on the Swiss CASCADE database. For Aim 3, feasibility and efficacy of the digital solution against the comparison intervention will be assessed in a randomized trial with a sample of 104 HBOC mutation carriers (52 in each arm). Aim 4 will be achieved with survey and interview data collected from HBOC families and healthcare providers during all phases of the study.

DETAILED DESCRIPTION:
The study will adapt and evaluate a digital platform to support communication of genetic test results in HBOC families. The Family Gene Toolkit (FGT) will be adapted to be less resource intensive and disseminated to a larger audience without increasing costs. The study will also develop the K-CASCADE research infrastructure in order to measure the long-term outcomes of the embedded randomized trial.

Methods

Aim 1: Develop a digital platform to support the communication of cancer predisposition among HBOC families, based on linguistic and cultural adaptation of the FGT for the Swiss and Korean population.

FGT included four modules designed to increase knowledge of cancer genetics (Module 1); provide decisional support for genetic testing (Module 2); increase active coping to common challenges faced by HBOC families (Module 3); provide a five-steps, skills-building communication training (Module 4). The digital health solution will be based on the four original modules and an additional fifth module, covering information about management of hereditary cancer risk based on the most updated national recommendations.

Team members will develop a custom web application to collect baseline information from participants, deliver the intervention and the comparator, randomize participants, collect follow up data, facilitate users to send text and email messages to relatives and share genetic testing results. Readily available e-learning products will create different tailored messages, multiple interactions and assessments, and an interface that can be accessed on desktop and mobile devices. Stakeholders will review the content online and provide feedback on word choices, sensitivity of messages, and appearance of the website. The Korean team will develop a module on cancer risk management options and the Swiss team will adapt and tailor the remaining modules.

The linguistic and cultural adaptation of FGT will be based on literature regarding implementation of health interventions and specific elements for message tailoring. The investigators will develop tailored messages in English and translate them into multilingual programs at the eighth grade reading level, taking into account social norms, legislation, health insurance policy, cultural values, and social networks.

Participants will be prompted to complete the five modules at their own pace within four weeks after they first engage with the intervention. The four-week interval will enable them to learn information in a sequential manner and to have adequate time to reflect and act based on the provided information, while also providing a controlled learning environment. Tailored feedback will be based on responses to questions in the baseline assessment. Within the four weeks, they will receive email alerts to visit the website and complete the five modules with the URL link that will direct them to the adapted FGT.

The comparison website will provide targeted information about HBOC and enable sharing genetic test results. The Korean team will define the contents of the comparator website that will mimic the structure and function of an existing website, and share a protocol for translations from English into Korean and Swiss languages.

Mini-focus groups with clinicians involved in genetic counseling will evaluate if the content of each module and the tailored messages are appropriate for the target populations. Focus groups with HBOC families will provide suggestions to enhance comprehensibility, usefulness, acceptability and feasibility of the intervention. Feedback received from clinicians and focus groups will help with further refinement of the content of each module and the tailored messages.

Usability and acceptability of a final version of the adapted FGT will be conducted with new members of the target population in each country. Participants will be asked to "think-aloud" while navigating the website and voice their thoughts, feelings, and opinions while they are completing each task. Usability testing will also help understand how to improve the interface. Feedback will be analyzed and incorporated into final revisions of the digital platform.

The Swiss sample will be identified through the five oncology and genetic testing centers participating in the CASCADE Consortium from three linguistic regions of Switzerland. The Korean sample will be identified from similar clinics in Seoul, Koyang, and Daejeon.

Focus groups with 20-24 participants (10-12 mutation carriers and 10-12 relatives) will be conducted at national language(s) of each country. There will be homogeneity within members of each focus group but the samples will be diversified in terms of demographics and clinical history between groups. Usability and acceptability testing will be performed with 5 new mutation carriers per country and language version.

Expert clinicians (6-10) involved in genetic consultation in each country and per linguistic region will be identified through the CASCADE Consortium and the SAKK Network in Switzerland, and through the KOHBRA network in Korea.

Recruitment for the focus groups will be done through the family-based cohort in Switzerland and/or flyers advertising the study posted in the affiliated institutions and clinics, and through social network service platforms in Korea. Focus groups will be co-lead by two members of the research team in each country, and each linguistic region in Switzerland. Usability testing sessions will be videotaped. Acceptability will be assessed with a seven-item survey assessing ease of use, clarity, appropriate length, level of detail, relevance, interest, and satisfaction.

Focus groups with HBOC families and clinicians will be audio recorded and transcribed verbatim, using codes to protect individual identification. Transcripts will be reviewed and content analyzed. Two members of the research team in each country will review the videotapes obtained from usability testing and the "think aloud" protocol. Data about usability and acceptability will be analyzed with descriptive statistics.

Aim 2: Develop the K-CASCADE research infrastructure in Korea by expanding an existing research infrastructure developed by the CASCADE Consortium in Switzerland

The design for K-CASCADE, assessments, and procedures for sample identification and data collection will follow procedures similar to the Swiss CASCADE study. The investigators will use this infrastructure to measure the long-term outcomes of the randomized trial.

Settings for recruitment will be open to interested member institutions within the KOHBRA network, with attention towards diversity in hospital geographical location and other characteristics to increase sample representativeness and generalizability. With an expected minimum of 5 hospital settings, over a period of 3 years, the accessible target population is estimated at 2,700 persons (15 persons/month x 12 months x 3 years x 5 hospitals), of which 50-60% roughly 1,350-1,600 individuals are estimated to participate. Korean men and women with an HBOC-associated pathogenic variant will be invited to participate and invite their first- and second-degree relatives, and their first cousins to the study. Investigators anticipate recruiting about 15 participants per month.

Mutation carriers identified in participating centers will be invited to the study with an invitation letter signed by their physician. Flyers will first be shared with clinicians via email and/or face-to-face meetings and patient advertisements will be posted in the centers.

For data collection on psychosocial variables, the Swiss CASCADE platform will be used to maintain consistency and accuracy of data entry, data cleaning and analyses. Korean respondents will be able to log on as K-CASCADE participants through the Swiss CASCADE website and participate in the baseline survey. For clinical data collection, written consent will be obtained from Korean participants who agree to share their health data, and their electronic medical records will be accessed and entered into a separate database by a Korean research associate.

Korean participants' data entered in the Swiss CASCADE platform will be available for descriptive and comparative analyses using their epidemiological and psychosocial data along with coded and non-identified clinical data.

Aim 3: Explore the benefits of the digital platform on psychological distress and communication of genetic test results, as well as knowledge of cancer genetics, coping, and decision making.

The investigators will assess the feasibility of delivering the intervention and indicators of engagement obtained from meta-data such as the number of modules accessed, time spent and the utilization of links, which are automatically recorded on the website. To assess intervention effects, a randomized controlled trial evaluating the adapted FGT compared to a comparison website will be conducted. Randomization will occur at the family level, i.e., the platform will randomly assign each mutation carrier and relatives to either intervention arm. Several instruments will be completed by all study participants at baseline (T1) prior to the intervention and again 2 months (T2) and 6 months (T3) later.

The Swiss sample will be identified through the oncology and genetic testing centers from three linguistic regions of Switzerland participating in the CASCADE Consortium. The Korean sample will be identified from similar clinics at Seoul, Koyang, and Daejeon.

The study will include 114 participants in order to have a total of N = 104 evaluable families (52 for each website). This sample size would allow detecting whether using the adapted FGT compared to the comparator website would increase the proportion of informed relatives by 25% with a statistical power of 80%, a significance level of 5%, and an expected drop-out rate of 9%. The investigators assumed an average of 2.8 relatives per family and the distribution of the proportion of relatives based on data from the Swiss family-based cohort.

The Swiss investigators anticipate identifying approximately 90 new mutation carriers per year from the five clinical centers affiliated with the CASCADE Consortium. In Korea, 150-250 new HBOC cases per year are estimated among the five participating institutions. From the pool of potential participants, it is expected that less than 10% have no relatives, and less than 10% have no access to a computer, tablet, or smartphone making them ineligible for the study. Based on similar studies it is expected that 75% of all eligible probands will participate in the study. Investigators expect to recruit and retain the necessary final sample of 114 individuals with an HBOC associated pathogenic variant and their relatives in about 18 months.

Potential participants carrying an HBOC-associated pathogenic variant will be emailed a code and the URL link to the website and a unique passcode to provide baseline assessments. To alleviate ethical concerns in contacting relatives without their explicit consent, mutation carriers will invite relatives to the website. By providing a signed consent, and completing the baseline survey, mutation carriers and relatives indicate their participation to the study. Eight weeks (T1) and six months (T2) after the first engagement with the intervention, participants will receive an email reminder to log in to the website and complete the follow up survey. Baseline and follow up surveys will each take about 30 minutes to complete.

Pre- and post-intervention data values from self-administered surveys will be checked for validity. Scales with alpha of 0.71 and higher will be used. Missing data will be dealt with multiple imputation or other techniques. The primary outcome will be calculated with a Wilcoxon-Mann-Whitney test to compare the proportions of informed relatives per study arm. Other primary and secondary data and metadata from automatic recording of website activity will be analyzed with descriptive statistics, including calculating means and frequencies of key variables and subject descriptors. Chi-square test for differences in proportions and t-test for differences in means will assess the associations between demographic factors and clinical characteristics. All analyses will be conducted using the statistical software R, using "two-sided" statistical tests and conﬁdence intervals with standard signiﬁcance and conﬁdence levels α = 5 % and (100 % - α) = 95 %.

Aim 4: Explore the reach, effectiveness, adoption, implementation, and maintenance of the digital platform.

To explore the potential for dissemination and implementation of the adapted FGT, the investigators will use the RE-AIM framework and explore reach, effectiveness, adoption, implementation, and maintenance of the adapted FGT at the individual and at the organizational level.

Information about the different dimensions of the RE-AIM framework will be collected with different formats, including refusal forms, study evaluation questions at the follow up survey, mini-interviews with non-participants and healthcare providers, and systematically collecting feedback from clinical settings about rates of cascade genetic testing in each country.

Data collected for Aim 4 will be analyzed with qualitative and quantitative methods presented in equivalent sections of Aim 1 and Aim 3. Narrative data obtained from mini-interviews will be audio recorded and transcribed verbatim, and analyzed for common themes. Descriptive analyses will include calculating means and frequencies of key variables and subject descriptors. Chi-square test for differences in proportions and T-test for differences in means will compare key variables between participants and non-participants.

ELIGIBILITY:
Inclusion Criteria:

* Speak and read German, French, Italian, English, or Korean
* Residence in Switzerland or in Korea
* Has been identified with a pathogenic variant associated with HBOC or
* Has ≥1 first-, second-degree relative or first cousing with HBOC
* Mentally able to provide informed consent

Exclusion Criteria:

* mutation carriers who do not have any family members;
* husbands and partners, although they may play an important role in decisions for genetic testing and risk management of disease, will not be included in the study;
* participants with a prior diagnosis of a mental disease and those unable to provide informed consent;
* those physically ill and not being able to complete a baseline survey;
* those without access to the web through a computer, tablet, or smartphone.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Profile of Mood States (POMS) | Baseline, 2 months and 6 months post-intervention
  Change in psychological distress of mutation carriers and relatives. The higher the score the higher the psychological distress.
Change in proportion of informed relatives | Baseline, 2 months and 6 months post-intervention
  Change in proportion of relatives that were invited to use the platform(s) over overall number of relatives eligible for cascade genetic testing
Informing Relatives Inventory | Baseline, 2 months and 6 months post-intervention
  Change in intention of mutation carriers to inform relatives about pathogenic variant and need for cascade genetic testing. The higher the score the higher the intention to inform relatives.
Intention to have genetic testing | Baseline, 2 months and 6 months post-intervention
  1 item, 7-point Likert-type scale ranging from 1 to 7 and assessing change in intention of untested, at risk relatives to have genetic testing. The higher the score the higher the intention to have genetic testing.
Reach | Baseline, 12 months, 24 months, 36 months, 48 months
  Change in the absolute number of individuals willing to participate in the study
Effectiveness | Baseline, 12 months, 24 months, 36 months, 48 months
  Change in number of "relative invites" initiated through the website
Adoption | Baseline, 12 months, 24 months, 36 months, 48 months
  Change in number of clinical sites willing to participate in the study
Implementation | Baseline, 12 months, 24 months, 36 months, 48 months
  Change in number of mutation carriers referred to the web-site
Maintenance | Baseline, 12 months, 24 months, 36 months, 48 months
  Change in number of visits to the web-site

SECONDARY OUTCOMES:
Acceptability - investigator developed | Baseline and 6 month post-intervention
  Change in attitude toward the intervention based on 16 items, 7 point Likert type scale. Minimum score 16, maximum 112, higher score indicates better acceptability
K-CASCADE | through study completion, an average of 4 years
  Number of individuals who take part in the study in Korea
Cancer diagnoses | Baseline, 12 months, 24 months, 36 months, 48 months
  Change in number of cancer diagnoses reported by participants
Cancer surveillance | Baseline, 12 months, 24 months, 36 months, 48 months
  Change in number of MRIs and mammograms reported by participants
Breast cancer risk factors and genetics knowledge index | Baseline, 2 month and 6 month post-intervention
  Change in genetic literacy and knowledge of genetic and epidemiological breast cancer risk factors. Minimum score 0, maximum score 36, higher score indicates higher knowledge of risk factors
Brief Cope | Baseline, 2 month and 6 month post-intervention
  Change in number of participants who engage in active coping e.g. information seeking vs. avoidance
Decision regret | Baseline, 2 month and 6 month post-intervention
  Change in decision regret for mutation carriers. Minimum score 5, maximum score 35, higher score means higher decision regret
Decision conflict | Baseline, 2 month and 6 month post-intervention
  Change in decision conflict for untested relatives. Minimum score 16, maximum score 112, higher score means higher decision conflict

CONTACTS AND LOCATIONS:
Overall Officials: Maria C. Katapodi, PhD, Principal Investigator — Department of Clinical Research, University of Basel
Locations (8):
- Switzerland (8):
  - HFR Fribourg - Hôpital cantonal, Fribourg, Canton of Fribourg
  - Hirslanden Clinic Des Grangettes, Geneva, Canton of Geneva
  - Hopital du Jura - Service d' Oncology, Delémont, Canton of Jura
  - Kantonalspital Winterthur, Winterthur, Canton of Zurich
  - University Hospital Basel, Basel
  - Istituto Oncologico della Zvizzera Italiana, Bellinzona
  - Universitatklinik fur Medizinische Onkologie, Inselspital, Bern
  - Unite d'Oncogenetique et de Prevention des Cancers, Geneva

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon completion of analyses addressing primary aims of the study - for 10 years
Access Criteria: Request protocol to CASCADE Consortium
URL: http://swisscascade.ch

REFERENCES:
- [Derived] Aceti M, Caiata-Zufferey M, Pedrazzani C, Schweighoffer R, Kim SY, Baroutsou V, Katapodi MC, Kim S; CASCADE and K-CASCADE Consortia. Modes of responsibility in disclosing cancer genetic test results to relatives: An analysis of Swiss and Korean narrative data. Patient Educ Couns. 2024 Jun;123:108202. doi: 10.1016/j.pec.2024.108202. Epub 2024 Feb 16. PMID 38395023
- [Derived] Kim S, Aceti M, Baroutsou V, Burki N, Caiata-Zufferey M, Cattaneo M, Chappuis PO, Ciorba FM, Graffeo-Galbiati R, Heinzelmann-Schwarz V, Jeong J, Jung MM, Kim SW, Kim J, Lim MC, Ming C, Monnerat C, Park HS, Park SH, Pedrazzani CA, Rabaglio M, Ryu JM, Saccilotto R, Wieser S, Zurrer-Hardi U, Katapodi MC. Using a Tailored Digital Health Intervention for Family Communication and Cascade Genetic Testing in Swiss and Korean Families With Hereditary Breast and Ovarian Cancer: Protocol for the DIALOGUE Study. JMIR Res Protoc. 2021 Jun 11;10(6):e26264. doi: 10.2196/26264. PMID 34114954